CLINICAL TRIAL: NCT06138535
Title: Evaluation of Digital Stabilizing Splint in Management of Masticatory Muscle Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: zahraa hassan (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor-Investigator, zahraa hassan, Principal Investigator, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZJD-D-23-00044
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Muscle Disorder
MeSH Terms: conditions — Muscular Diseases | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: single arm group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Masticatory Muscle Disorder patients treated by digital stabilizing splint (Other): digital stabilizing splint
  Interventions: Device: digital stabilizing splint

INTERVENTIONS:
Device: digital stabilizing splint — 3D Printed stabilizing splint that has been digitally designed on a modern software
  Other Names: occlusal splint

SUMMARY:
The goal of this clinical trial is to evaluate the digital stabilizing splint in management of masticatory muscle disorder. The main question it aims to answer are:

• is the digital stabilizing splint effective in treatment of masticatory muscle disorder signs and symptoms after 3 months follow up ? Participants will be asked to ware the splint and progressively increasing the duration of splint wear, starting from 8 hours per day for 3 months .

DETAILED DESCRIPTION:
The current research was conducted for evaluation of the digital stabilizing splint in the management of masticatory muscle disorder. Subjects and Methods: Eight patients over the age of 18 with masticatory muscle disorders received treatment using a stabilizing splint that was digitally created. The Each patient's response to therapy modifications was assessed and compared before and after splint insertion for each patient subjective symptoms were assessed using a patient questionnaire that was repeated before treatment (baseline), one month, and 3 months post-insertion. Moreover, The masseter and temporalis muscles' electrical activity was measured using electromyography at baseline and after three months.post-splint insertion. Clinical signs such as mouth-opening lateral movements and protrusive movements were measured before and 3 months after the splint was inserted.

ELIGIBILITY:
inclusion criteria

1-Anterior disc displacement without reduction or osteoarthritis cases 2-Pain and/or tenderness of masticatory muscles exclusion criteria

1. Absence of previous occlusal splint therapy.
2. Absence of apparent dental or periodontal diseases.
3. Patients having full or partial dentures that would compromise the support of an occlusal splint were excluded.
4. Patient taking analgesics, muscle relaxants, or Anti-inflammatory medications will not be included because they may affect the outcome.
5. Patients with multiple teeth loss that affects occlusal splint support were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Patient questionnaire (clinical symptoms). | 3 months
  Patient questionnaire (clinical symptoms) . The questionnaire was used to detect the clinical symptoms scoring that ranges from 0 to 10 (10 being greatest pain/dysfunction and 0 signifying no pain/proper function).
  The success or failure was determined by the reduction in pain and dysfunction postoperatively.
  the scales were taken for all eight patients before and after 3 months of treatment.
  the questionnaire included questions about different clinical symptoms as following: headaches, facial discomfort, jaw joint pain, pain during mastication, neck pain, difficulty opening the mouth, difficulty in jaw movements, complaints during chewing, and clenching habits.

SECONDARY OUTCOMES:
Clinical sign such as mouth opening | 3 months
  Clinical sign such as mouth opening that was recorded by measuring the distance between the upper and lower central incisors by a caliper in millimeters unit.
  the increase in mouth opening indicates positive clinical improvement. the mouth opening was measured before and after 3 months of treatment.

OTHER OUTCOMES:
Evaluation of muscle activation with surface electromyography (EMG) | 3 months
  Evaluation of muscle activation with surface electromyography (EMG) for each of the eight patients enrolled in our study, and the records were taken before and after 3 months of treatment.
  The surface electrodes were placed on the anterior temporalis and the superficial masseter muscles.
  A Fast Fourier Transform ( FFT ) was carried out using the software of electromyography. The mean value of the EMG activity of each muscle was calculated from the amplitude in microvolts ( μV ).
  The decrease in the muscle records was an indication of improvement of muscle activity.

CONTACTS AND LOCATIONS:
Overall Officials: zahraa hassan, Principal Investigator — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data may be obtained either from study investigators or via data-sharing repositories or platforms.
Supporting Information: ICF
Time Frame: one yaer
Access Criteria: Al-Azhar Journal of Dentistry
URL: https://azjd.researchcommons.org/